CLINICAL TRIAL: NCT05940207
Title: Safety Testing of Hydrogen Peroxide-Generating e-Bandage on Normal Human Skin
Brief Title: A Study of Hydrogen Peroxide-Generating E-bandage Safety
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Principal Investigator, Robin Patel, Principal Investigator, Mayo Clinic
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Other
Other Study IDs: 23-003805
Record Dates: First submitted 2023-07-03; First posted 2023-07-11 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2026-01

CONDITIONS: Healthy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (5):
- e-Bandages 3 hours (Experimental): Four subjects will wear the e-Bandage on their skin for 24 hours, with active polarization for 3 hours.
  Interventions: Device: e-Bandages
- e-Bandages 6 hours (Experimental): Four subjects will wear the e-Bandage on their skin for 24 hours, with active polarization for 6 hours.
  Interventions: Device: e-Bandages
- e-Bandages 12 hours (Experimental): Four subjects will wear the e-Bandage on their skin for 24 hours, with active polarization for 12 hours.
  Interventions: Device: e-Bandages
- e-Bandages 24 hours (Experimental): Four subjects will wear the e-Bandage on their skin for 24 hours, with active polarization for 24 hours.
  Interventions: Device: e-Bandages
- Control Group (Experimental): Four subjects will wear the e-Bandage on their skin for 24 hours, with no active polarization.
  Interventions: Device: e-Bandages

INTERVENTIONS:
Device: e-Bandages — A hydrogen-peroxide generating e-bandage for wound infection and treatment and prevention. Each e-bandage is composed of three electrodes - a working, a counter, and a reference electrode. Cotton fabric physically separates electrodes. Constant (regulated) generation of low-concentrations of hydrogen peroxide happens on the working electrode, which is in contact with the skin covered with a hydrogel layer.

SUMMARY:
A novel hydrogen peroxide-generating electrochemical bandage for wound infection treatment and prevention, and wound healing has been developed. The purpose of this research is to gather information on the safety and to confirm lack of toxicity of small hydrogen peroxide-generating e-bandages on normal human skin.

ELIGIBILITY:
Inclusion Criteria:

* Healthy.
* Intact skin on arms.
* Able to provide appropriate consent.

Exclusion Criteria:

* Vulnerable study population.
* Pregnancy.
* Children.
* Skin disease.
* Non-intact skin on arms.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-03-27 (Actual); Primary Completion 2029-05 (Estimated); Study Completion 2029-05 (Estimated)

PRIMARY OUTCOMES:
e-Bandage Discomfort | Approximately 3 - 24 hours
  Self-report discomfort with the e-Bandage, graded on a scale of 1-4, with 1 being no reaction, 2 mild reaction, 3 moderate reaction, 4 severe reaction.
Skin irritation/dermatitis | Approximately 3 - 24 hours
  Skin redness or swelling, graded on a scale of 1-4, with 1 being no reaction, 2 mild reaction, 3 moderate reaction, 4 severe reaction.
Allergic Reaction | Approximately 3 - 24 hours
  Local/systemic allergic reaction to the e-Bandage, graded on a scale of 1-4, with 1 being no reaction, 2 mild reaction, 3 moderate reaction, 4 severe reaction.
Skin Discoloration | Approximately 3 - 24 hours
  Skin discoloration from the e-Bandage, graded on a scale of 1-4, with 1 being no reaction, 2 mild reaction, 3 moderate reaction, 4 severe reaction.

CONTACTS AND LOCATIONS:
Overall Officials: Robin Patel, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic Minnesota, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kies PJ, Kim WJ, Fleming D, Bozyel I, Holtegaard S, Shrivastava S, Schwartz K, Schwieder S, Beyenal H, Patel R. Safety trial assessing 1.77 cm2 H2O2 producing electrochemical bandages on healthy human skin. Sci Rep. 2025 Oct 30;15(1):38074. doi: 10.1038/s41598-025-21803-y. PMID 41168214